CLINICAL TRIAL: NCT05711433
Title: Risk Factors for Postoperative Pancreatic Fistula Following Non-traumatic Pancreatic Surgery. Retrospective Observational Study.
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, assistant professour of general and laparoscopic surgery, Zagazig University
Other Study IDs: zagazig 16
Record Dates: First submitted 2022-10-21; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Pancreas Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 42 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pancreatic surgery — pancreaticoduodenectomy and distal pancreatectomy

SUMMARY:
Postoperative pancreatic fistula is a potentially fatal sequela with substantial morbidity and mortality. A retrospective observational study was conducted in the surgical unit of Zagazig university hospital . Three hundred forty-seven patients were admitted with a clinical diagnosis of pancreatic fistula following both open and laparoscopic approaches for pancreatic benign and malignant tumors.

DETAILED DESCRIPTION:
Postoperative pancreatic fistula is a potentially fatal sequela with substantial morbidity and mortality. POPF incidence and risk factors vary.

A retrospective observational study was conducted in the surgical unit of Zagazig university hospital . Three hundred forty-seven patients were admitted with a clinical diagnosis of pancreatic fistula following both open and laparoscopic approaches for pancreatic benign and malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years,
* both sexes,
* respectablee pancreaticoduodenal tumors, or chronic pancreatitis

Exclusion Criteria:

* <18 years,
* Patients who underwent total pancreatectomies,
* Patients discovered intraoperatively to be fixed to portal vein or superior mesenteric artery, traumatic pancreatic surgeries, postoperative associated gastric or biliary leak, pancreaticoduodenal cancers infiltrating the colon, stomach or liver.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A retrospective observational study was conducted in the surgical unit of Zagazig university hospital from July 2014 to July 2019. Three hundred forty-seven patients were admitted with a clinical diagnosis of pancreatic fistula following both open and laparoscopic approaches for pancreatic benign and malignant tumors.
Sampling Method: Non-Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative pancreatic fistula | 3.5 years
  an amylase level in the fluid collected from the drain on the third postoperative day (POD) that was > three times the serum amylase level

IPD SHARING:
Plan to Share IPD: No